CLINICAL TRIAL: NCT06671418
Title: Primary Percutaneous Stenting Above the Ampulla Versus Endoscopic Drainage for Unresectable Malignant Hilar Biliary Obstruction (TESLA RCT)
Brief Title: Primary Percutaneous Stenting Above the Ampulla Versus Endoscopic Drainage for Unresectable Malignant Hilar Biliary Obstruction
Acronym: TESLA RCT
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Bas Groot Koerkamp, MD, PhD, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Erasmus MC TESLA RCT
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Cholangiocarcinoma Non-resectable; Gall Bladder Cancer; Liver Metastasis; Malignant Hilar Stricture
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopic biliary drainage (standard of care) (Other)
  Interventions: Procedure: Endoscopic biliary drainage
- Primary percutaneous stenting (Active Comparator)
  Interventions: Procedure: Primary percutaneous stenting (PPS)

INTERVENTIONS:
Procedure: Primary percutaneous stenting (PPS) — PPS bridging malignant hilar biliary obstruction with self-expandable uncovered metal stents without crossing the ampulla and without leaving an external drain. The procedure is performed by an interventional radiologist who has performed at least 5 PPS procedures.
  Arms: Primary percutaneous stenting
Procedure: Endoscopic biliary drainage — EBD according to the American Society for Gastrointestinal Endoscopy (ASGE) guidelines of 2021. The procedure is performed by a gastro-enterologist who is experienced in performing EBD in patients with a MHBO.
  Arms: Endoscopic biliary drainage (standard of care)

SUMMARY:
The goal of this clinical randomized controlled trial is to perform primary percutaneous stenting (PPS) in patients with malignant hilar biliary obstruction (MHBO). The main question it aims to answer is:

To compare the efficacy of PPS above the ampulla to standard endoscopic biliary drainage (EBD) in patients with a MHBO who are ineligible for surgical resection.

Researchers will compare PPS with EBD to see if major complications within 90 days after randomisation occur.

Participants will undergo either primary percutaneous stenting or endoscopic biliary drainage, depending on randomization.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be given according to ICH/GCP and national/local regulations.
* MHBO on imaging with histopathological confirmation or high clinical suspicion.
* Ineligible for surgical resection.
* Hyperbilirubinemia (a combination of a total bilirubin level >50 mmol/l.

Exclusion Criteria:

* Fluctuation or spontaneous decrease of a total bilirubin level before start of any treatment suggesting a potential non-malignant diagnosis.
* Patients who underwent previous biliary drainage procedures endoscopically or percutaneously. Patients who underwent an attempted but failed ERCP are eligible only when no papillotomy or cannulation was performed.
* Clinical signs of cholangitis. Cholangitis is defined as the presence of both fever (i.e. body temperature >38.5°C) and leucocytosis (i.e. ≥10 *109/L) without clinical or radiological evidence of acute cholecystitis (22).
* Uncorrectable coagulation disorder.
* Uncorrectable contrast allergy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Major complications within 90 days after randomisation | 90 days after randomization
  The primary objective is to compare major complications within 90 days after randomization of PPS and EBD in patients with MHBO who are ineligible for surgical resection. Major complications are defined as any complication leading to prolonged hospital stay of more than 72 hours, readmission to hospital, invasive reintervention, or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rousian M, van Verschuer V, Franssen S, Bijdevaate D, Bokkers RPH, Braat AE, de Bruijne J, Bruno MJ, Burgmans MC, van Delden OM, Dewulf M, Erdmann JI, Hagendoorn J, van der Holt B, Hoogwater FJH, Inderson A, van der Leij C, Mohseny B, Poley JW, Smits MLJ, van Vilsteren FGI, Voermans RP, Zijlstra IAJ, van Driel LMJW, Koerkamp BG. Primary percutaneous stenting above the ampulla versus endoscopic drainage for unresectable malignant hilar biliary obstruction (TESLA RCT): study protocol for a multicenter randomized controlled trial. BMC Cancer. 2025 May 9;25(1):849. doi: 10.1186/s12885-025-14158-0. PMID 40346549